CLINICAL TRIAL: NCT02425787
Title: The Bereaved Parent Study
Brief Title: Bereaved Parent Study
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BPS14
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Bereavement
Keywords: Loss of a child; Grief
MeSH Terms: interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Parents of deceased children (no BMT): Participants will be parents who have lost a child at St. Jude Children's Research Hospital (SJCRH). They will participate in a 60-90 minute interview.
  (Not recruiting)
  Interventions: Behavioral: Interview
- Parents of deceased children (haploidentical BMT): Participants will be parents whose child died after receiving a haploidentical bone marrow transplant at St. Jude Children's Research Hospital (SJCRH), and who have not previously participated in an interview through this study. They will participate in a 30-90 minute interview.
  Interventions: Behavioral: Interview
- Parents of deceased children (non-haploidentical BMT): Participants will be parents whose child died after receiving a non-haploidentical bone marrow transplant at St. Jude Children's Research Hospital (SJCRH), and who have not previously participated in an interview through this study. They will participate in a 30-90 minute interview.
  Interventions: Behavioral: Interview
- Parents of deceased children (not interviewed): Participants will be parents who have lost a child at SJCRH, who have not previously participated in an interview through this study.They will participate in a 30-90 minute focus group.
  Interventions: Behavioral: Focus Group
- Hematology/Oncology Fellows: Participants will be Hematology/Oncology Fellows at SJCRH. They will participate in a 30-90 minute focus group.
  Interventions: Behavioral: Focus Group
- Legacy-Building: Participants will be parents who have lost a child at SJCRH and received legacy items. They will participate in a 30-90 minute interview.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — This is a prospective study with a semi-structured in-depth qualitative interview. Interviews will be conducted by the study PI or designee. However, in order to ensure that the interviews are conducted sensitively, the first 10 interviews will be observed and supervised by a clinically credentialed St. Jude faculty member, and an additional 10% of the interviews will be observed after that.
  In order to ensure that the interviewer does not lead the participant, or in turn, that the participant does not feel limited in regards to what they believe is an appropriate or desired response, the semi-structured interview questions are general and intended to produce broad responses in regards to participant experiences.
  Other Names: Questions
  Groups: Parents of deceased children (haploidentical BMT); Parents of deceased children (no BMT); Parents of deceased children (non-haploidentical BMT)
Behavioral: Focus Group — Focus groups will be conducted with a two-fold purpose in mind:
  1. With bereaved parents: to validate the findings of the preliminary analyses of the initial interviews &/or to suggest avenues of further inquiry to expand and more deeply define the grief journey of bereaved parents.
  2. With Hematology/Oncology Fellows: to receive input regarding the applicability and use of the findings during the training and future careers of these medical providers.
  Other Names: Group question/answer sessions
  Groups: Hematology/Oncology Fellows; Parents of deceased children (not interviewed)
Behavioral: Interview — The interview will be conducted by study team members and will center around legacy item-related questions.
  Other Names: Questions
  Groups: Legacy-Building

SUMMARY:
Recent focus groups at St. Jude Children's Research Hospital (SJCRH) revealed several limitations in our understanding of how parents' relationships with care staff help and hinder their grief experience. Additionally, there is a gap in the bereavement literature regarding the psychological effects professional caregiver relationships have on parents whose children died of cancer. To bolster our knowledge base and benefit Bereavement Care Services at SJCRH, as well as benefit other professionals by filling the gap in the literature, we have designed a qualitative study that will conduct individual interviews with bereaved parents whose children died at SJCRH.

Validation of the preliminary analyses of the initial 30 interviews will occur through new focus groups involving two separate sets of bereaved parents who will validate the findings and/or suggest additional avenues of inquiry needed to gain a more complete understanding of parental grief/bereavement experience. Additionally, focus groups with hematology/oncology fellows will obtain provider feedback on the value of these findings in their training and future role as physicians.

The initial focus group portion of this study is complete and more than 30 interviews have been conducted with bereaved parent participants. Review of those interviews revealed that very few parent participants had children who received bone marrow transplants. For this reason, we will now specifically be recruiting bereaved parent participants whose children received bone marrow transplants at St. Jude Children's Research Hospital. We will be recruiting parents of children who received haploidentical and non-haploidentical bone marrow transplants because we believe the parents of deceased children who received haploidentical bone marrow transplants may have unique bereavement experiences related to their possible roles as donors. The act of donating or not being selected to donate to a child who goes on to die from cancer and its related complications may have unique impacts on the grieving process and warrants specific investigation. We also hope to better understand how legacy building interventions are perceived and utilized by caregivers following the death of a child from cancer.

DETAILED DESCRIPTION:
Participants who consent will engage with the principal investigator in a one-time voice-recorded interview consisting of demographic and open-ended questions. Participants can choose to conduct the interview face-to-face or over-the-phone. Completion of the interview is expected to take between 30-90 minutes. Validation focus groups are expected to take between 30-90 minutes, as well. For the legacy-building cohort, the Child Life Department will provide additional information to specify which bereaved families received legacy items, and parents will be recruited to participate in an interview centered on the legacy item questions.

PRIMARY OBJECTIVE

To conduct qualitative interviews in order to understand what helps and what hinders bereavement processes among St. Jude parents, with particular attention to how relationships with St. Jude professional care staff affect parental bereavement processes.

EXPLORATORY OBJECTIVES

To qualitatively explore the unique bereavement experiences and challenges of parents of children who have received bone marrow transplantation, and compare these experiences with those participants whose children did not receive bone marrow transplantation.

To assess for qualitative similarities among parents with similar responses on questionnaires and/or to identify between-group differences on questionnaires among parents with qualitatively similar experiences.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* Must be English-speaking.
* Must have had a child who received oncological treatment at SJCRH.
* The child who received treatment must have died at least 1 year prior but no more than 6 years ago, with the cause of death related to progressive cancer or cancer-related complications.

OR

* English-speaking Hematology/oncology Fellows at SJCRH who are at least 17 years of age.

Exclusion Criteria:

* Potential participants who indicate active suicidal ideation with or without plans will be excluded from the study. Appropriate care and referral will be given as indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents who have lost a child at SJCRH and who consent to participate in the individual interviews or follow-up focus groups. Hematology/oncology Fellows at SJCRH who consent to participate in the follow up focus groups..
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Descriptive accounts of bereavement | Once, Day 0
  Qualitative data will be collected using a standardized semi-structured interview technique. Researchers will analyze transcripts for content to gain a better understanding of the bereavement experience. Thematic saturation will occur when a minimum of 3 consecutive interviews fail to produce novel information in each of the therapeutic categories (haploidentical transplant, non-haploidentical transplant).Transcripts will be analyzed as they are obtained and the principal investigator and study team will iteratively and collaboratively develop a coding dictionary. Each transcript will be reviewed by at least 2 coders. When there is disagreement on a code, coders will meet in person to discuss until consensus is reached. Codes will be grouped into broader themes and used to summarize and describe the bereavement experience as told by parents.

OTHER OUTCOMES:
To qualitatively explore the unique bereavement experiences and challenges of parents of children who received bone marrow transplantation, and compare these experiences with those participants whose children did not receive bone marrow transplantation. | All data will be collected at the time of the initial interview.
  We will use qualitative content analysis as described above to identify similarities and differences among the different cohorts of bereaved parents (parents whose children did not receive bone marrow transplantation, parents whose children received haploidentical bone marrow transplantation, and parents whose children received non-haploidentical bone marrow transplantation.
To assess for qualitative similarities among parents with similar responses on questionnaires and/or to identify between-group differences on questionnaires among parents with qualitatively similar experiences. | All data will be collected at the time of the initial interview.
  We will use the Beck Depression Inventory-II (BDI-II) to assess for symptoms of depression, the parental grief disorder questionnaire (PG-13) to assess for atypical or disordered grief, and the Integration of Stressful Life Experiences Scales (ISLES-SF) to measure the extent to which the child's loss has been integrated into the parent's worldview. We will identify different groups based on these questionnaires (ex: those with elevated scores on the BDI-II) and look to see if the thematic content of their interviews differs from other participants. Additionally, we may identify participants who expressed certain themes and assess for differences in their qualitative responses.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Baker, MD, Principal Investigator — St. Jude Children's Research Hospital; Erica C. Kaye, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols